CLINICAL TRIAL: NCT04276922
Title: Creative Arts Program to Reduce Burnout in Healthcare Professionals
Acronym: CORAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2759; NEAPS1801 (Other Grant/Funding Number: National Endowment for the Arts)
Record Dates: First submitted 2020-01-30; First posted 2020-02-19 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Burn-Out Syndrome; Post-Traumatic Stress Disorder; Depression, Anxiety
MeSH Terms: conditions — Burnout, Psychological; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders | interventions — Music Therapy; Movement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Visual Arts Group (Experimental): Visual Arts group - sketch journals
  Interventions: Behavioral: Visual Arts
- Music Group (Experimental): Music group involves music-listening exercises (such as lyric analysis, patient-chosen, music for relaxation and/or visualization) and active music making.
  Interventions: Behavioral: Music
- Dance/Movement Group (Experimental): Dance/Movement group - movement check-in, gentle physical warm-up, and then either a structured or improvisational movement process.
  Interventions: Behavioral: Dance/Movement
- Writing/Poetry Group (Experimental): Writing/Poetry group uses writing workshops using integral elements of good writing.
  Interventions: Behavioral: Writing/Poetry
- Control Group (Experimental): Surveys at baseline and 12 weeks later.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Visual Arts — Subjects meet for 90 minutes, once weekly, over 12 weeks for guided drawing/sketching sessions. The 12 sessions will follow a standard sequence that addresses three primary themes: creating safety, inviting vulnerability, and integrating into a transformative community.
  Surveys, activity diary cards will be completed at baseline, weekly and at intervention completion to assess satisfaction, stress, and well-being. Qualitative focus groups will occur after the intervention to assess acceptability of intervention, outcomes assessments, program development and implementation.
  Arms: Visual Arts Group
Behavioral: Music — Subjects meet for 90 minutes, once weekly, over 12 weeks, for guided music-listening exercises (such as lyric analysis, patient-chosen, music for relaxation and/or visualization) and active music making. The 12 sessions follow a standard sequence, addressing three primary themes: creating safety, inviting vulnerability, and integrating into a transformative community.
  Surveys, activity diary cards are completed at baseline, weekly and at completion to assess satisfaction, stress, and well-being. Qualitative focus groups, after the intervention, assess acceptability of intervention, outcomes, program development and implementation.
  Arms: Music Group
Behavioral: Dance/Movement — Subjects will meet once weekly, and begin with a movement check-in, a gentle physical warm-up, and then either a structured or improvisational movement process. for a total of 12 weeks. Each session will last 90 minutes. The 12 sessions will follow a standard sequence that addresses three primary themes: creating safety, inviting vulnerability, and integrating into a transformative community.
  Surveys, activity diary cards will be completed at baseline, weekly and at intervention completion to assess satisfaction, stress, and well-being. Qualitative focus groups will occur after the intervention to assess acceptability of intervention, outcomes assessments, program development and implementation.
  Arms: Dance/Movement Group
Behavioral: Writing/Poetry — Subjects will meet once weekly, for writing workshops to encourage participants to tell the stories they need to tell, using integral elements of good writing, for a total of 12 weeks. Each session will last 90 minutes. The 12 sessions will follow a standard sequence that addresses three primary themes: creating safety, inviting vulnerability, and integrating into a transformative community.
  Surveys, activity diary cards will be completed at baseline, weekly and at intervention completion to assess satisfaction, stress, and well-being. Qualitative focus groups will occur after the intervention to assess acceptability of intervention, outcomes assessments, program development and implementation.
  Arms: Writing/Poetry Group
Behavioral: Control — Control Group will only complete surveys at baseline and 12 weeks later.
  Arms: Control Group

SUMMARY:
This study plans to learn if creative arts programs that include visual, musical, written, or physical expression can reduce symptoms of burnout syndrome, Post Traumatic Stress Disorder (PTSD), depression, and anxiety in critical care healthcare professionals. This study also explores if creative arts can enhance the connection to the purpose of work, the development of adequate coping skills, while providing time to connect with peers.

ELIGIBILITY:
Inclusion Criteria:

* Employed as a healthcare provider, practicing primarily in a hospital setting for at least 20 hours per week.
* Positive symptoms of burnout measured via the Maslach Burnout Inventory (MBI):

  * emotional exhaustion score of >17, or
  * depersonalization score of >7, or
  * personal accomplishment score of < 31.

Exclusion Criteria:

• Unwillingness to participate in any of the four creative arts interventions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability/Satisfaction of Intervention as assessed by Client Satisfaction Questionnaire (CSQ-8) scores to yield a homogeneous estimate of general satisfaction. | At the end of 12 week intervention
  Acceptability of intervention will be assessed using eight item Client Satisfaction Questionnaire (SCQ-8) to generate an estimate of general satisfaction. Scores range from 8-32 (higher scores = greater satisfaction).

SECONDARY OUTCOMES:
Change in subject perception of intervention process scores as assessed by Psychological General Well-Being Index (PGWBI). | Baseline and after 12 weeks
  Emotional experience and sense of achievement using Psychological General Well-Being Index (PGWB), uses a 22-item survey to produce a single measure of psychological well-being.
Change in subject perception of intervention process scores as assessed by Positive and Negative Affect Schedule (PANAS). | Baseline and after 12 weeks
  Positive and Negative Affect Schedule (PANAS) is a 20-item, self-report measure for changes in mood. Positive and negative affect (PA/NA) reflect dispositional dimensions - high-NA reflects subjective distress and unpleasable engagement, while high-PA represents pleasurable engagement, such as enthusiasm and alertness; low-PA reflects lethargy and sadness.
Change in subject perception of intervention process scores as assessed by Maugeri Stress Index (MASI). | Baseline and after 12 weeks
  Maugeri Stress Index (MASI) is a self-report questionnaire. Four correlated sub scales (Wellness, Resilience, Perception of social support, and Negative coping styles). Total index is sum of responses (coded from 1 to 5). MASI-R score is expressed as a continuous variable: range: 0-100 , 50th percentile or less indicates presence of a stress condition) 118.
Change in perceived occupational stress as assessed by Medical Personnel Stress Survey (MPSS-R). | Baseline and after 12 weeks
  Medical Personnel Stress Survey (MPSS-R) assesses key stressors on organizational and individual levels. Measures 4 components of occupational stress: organizational stress, job dissatisfaction, negative patient attitudes, somatic distress.
Change in perceived occupational stress as assessed by Job Content Questionnaire (JCQ). | Baseline and after 12 weeks
  Job Content Questionnaire (JCQ) is scored on a 4-point Likert scale, covers 3 dimensions: Psychological Demand: 9 items evaluating amount of work demanded, rapidity required, time available, and level of concentration required. Decision Latitude: 9 items evaluating decision authority, use of skills, and varied aspects of tasks. Social support: 8 items evaluating help and interest provided by colleagues and supervisors.
Change in perceived occupational stress as assessed by Turnover Intention Questionnaire (TIQ). | Baseline and after 12 weeks
  Turnover Intention Questionnaire (TIQ): 6 single-choice questions asking the respondents' intention to leave. Responses scored 1-4. High scores indicate high intention level to leave the profession. Total score of turnover intention is divided into four levels: lower ≤6, low >6 and ≤12, high >12 and ≤18, higher>18.
Change in level of psychological distress as measured by Posttraumatic Diagnostic Scale (PDS). | Baseline and after 12 weeks
  Posttraumatic Diagnostic Scale (PDS) yields both a DSM-V diagnosis and symptom severity. Calculated by having a traumatic event, and a re-experiencing criterion, three avoidance symptoms, and two arousal symptoms.
Change in level of psychological distress as measured by the Hospital Anxiety Depression Scale (HADS). | Baseline and after 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) assesses 7-item anxiety subscale and a 7-item depression subscale. A score of > 8 identifies a positive history of anxiety or depression symptoms.
Change in level of Burnout as measured by Maslach Burnout Inventory. | Baseline and after 12 weeks.
  Maslach Burnout Inventory: Collected at baseline and post intervention.
  Maslach Burnout Inventory (MBI) designates positive symptoms of burnout via three areas: emotional exhaustion score of >17, depersonalization score of >7, or a personal accomplishment score of < 31.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Moss M, Edelblute A, Sinn H, Torres K, Forster J, Adams T, Morgan C, Henry M, Reed K. The Effect of Creative Arts Therapy on Psychological Distress in Health Care Professionals. Am J Med. 2022 Oct;135(10):1255-1262.e5. doi: 10.1016/j.amjmed.2022.04.016. Epub 2022 May 14. PMID 35576997